CLINICAL TRIAL: NCT02150824
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Groups Study to Investigate the Safety and Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of Three BI 187004 Doses Given Once Daily as Mono-therapy and of the Highest BI 187004 Dose Given Once Daily as Add on Treatment to Metformin Over 28 Days in Patients With Type 2 Diabetes Mellitus
Brief Title: Safety and Tolerability, Efficacy, Pharmacokinetic and Pharmacodynamic Study of Three Doses of BI 187004 Over 28 Days in Patients With Type 2 Diabetes Mellitus With and Without Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1307.4; 2013-003646-16 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (4):
- BI 187004 low dose mono QD (Experimental): patient to receive one tablet containing low dose of BI 187004 or matching placebo
  Interventions: Drug: Placebo; Drug: BI 187004
- BI 187004 medium dose mono QD (Experimental): patient to receive one tablet containing medium dose mg of BI 187004 or matching placebo
  Interventions: Drug: Placebo; Drug: BI 187004
- BI 187004 high dose mono QD (Experimental): patient to receive one tablet containing high dose of BI 187004 or matching placebo
  Interventions: Drug: Placebo; Drug: BI 187004
- BI 187004 high dose QD add on (Experimental): patient to receive one tablet containing high dose of BI 187004 or matching placebo add on to metformin background dose
  Interventions: Drug: Placebo; Drug: BI 187004

INTERVENTIONS:
Drug: Placebo — BI 187004 high dose matching placebo once daily
  Arms: BI 187004 high dose mono QD
Drug: Placebo — BI 187004 medium dose matching placebo once daily
  Arms: BI 187004 medium dose mono QD
Drug: Placebo — BI 187004 high dose matching placebo once daily add on to background metformin
  Arms: BI 187004 high dose QD add on
Drug: BI 187004 — BI 187004 high dose once daily add on to background metformin
  Arms: BI 187004 high dose QD add on
Drug: Placebo — BI 187004 low dose matching placebo once daily
  Arms: BI 187004 low dose mono QD
Drug: BI 187004 — BI 187004 medium dose once daily
  Arms: BI 187004 medium dose mono QD
Drug: BI 187004 — BI 187004 low dose once daily
  Arms: BI 187004 low dose mono QD
Drug: BI 187004 — BI 187004 high dose once daily
  Arms: BI 187004 high dose mono QD

SUMMARY:
Assess the safety and tolerability of once daily oral doses of BI 187004 in patients with type 2 diabetes mellitus without oral antidiabetic treatment and in patients on a stable metformin background treatment over 28 days. Assess the effect on fasting plasma glucose after 28 days of treatment and to investigate the pharmacokinetics and pharmacodynamics of BI 187004.

ELIGIBILITY:
Inclusion criteria:

1. Male or postmenopausal or hysterectomised female patients with diagnosis of Type 2 Diabetes Mellitus (T2DM) before informed consent
2. To be eligible for Arm 1

   1. Oral antidiabetic mono-therapy for the last 12 weeks prior to Informed Consent AND Glycosylated haemoglobin (HbA1c) >= 6.5% and <= 8.5% at Visit 1a
   2. Therapy-naïve patients or no antidiabetic treatment within 4 weeks prior to Informed Consent AND HbA1c >= 7.0% and <= 9.5% at Visit 1a.
3. To be eligible for Arm 2:

   a. Antidiabetic treatment with metformin with an unchanged daily dose for 12 weeks prior to Informed Consent AND patient´s willingness to keep this therapy stable during the course of the trial AND HbA1c >= 7.0% and <= 9.5% at Visit 1a
4. Age >=18 and <=80 years for female hysterectomised and male patients at Visit 1a
5. Age >=55 and <=80 years for female postmenopausal (defined by the absence of menses for at least 2 years) patients at Visit 1a
6. Body mass index (BMI) >= 28 and <= 40 kg/m2 at Visit 1a
7. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion criteria:

1. Treatment with a non-oral antidiabetic therapy or with more than one oral antidiabetic medication within 12 weeks prior to visit 1a.
2. Fasted plasma glucose > 240 mg/dl (>13.3 mmol/l) on two consecutive days after screening (Visit 1a) confirmed by a fasted laboratory blood glucose test until first administration of the trial drug
3. Any laboratory value more than 3 times above upper limit normal (ULN) at screening (visit 1a) or any other laboratory value outside the reference range and clinically relevant in the investigator judgment
4. Any known clinically relevant concomitant diseases or chronic diseases other than type 2 diabetes, hyperlipidaemia or medically treated hypertension
5. Medical history of cancer or treatment for cancer in the last five years prior to the Visit 1a.
6. History of Cushing syndrome, Addison´s disease, congenital adrenal hyperplasia or polycystic ovary syndrome
7. Treatment with systemic, inhalatory or ophthalmologic steroids within 12 weeks prior to first administration of the trial drug.
8. Treatment compliance during the run-in period is outside the per protocol range defined range, between 80%-120% treatment compliance.
9. Use of any other concomitant medication within 5 half-lives before the first administration of the trial drug except for allowed co-medication.
10. Surgery or trauma with significant blood loss (more than 500 ml) within the last 3 months prior to informed consent or blood donation (more than 100 ml) within four weeks prior to first administration of study medication or planned during the trial
11. Any other medical condition that would interfere with trial participation based on investigator´s judgement or any on-going clinical condition that would jeopardize patient´s or site personnel´s safety or study compliance based on investigator judgement. Smoking habits interfering with hospitalization. Patients not willing to abstain from alcoholic beverages during inpatient visits
12. Male patients not willing to use adequate contraception (sexual abstinence, condom use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the whole study period from the time of the first intake of study drug until three months after the last intake

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with drug- related adverse events | 6 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose (FPG) after 28 days of treatment | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Germany (3):
  - 1307.4.49003 Boehringer Ingelheim Investigational Site, Berlin
  - 1307.4.49002 Boehringer Ingelheim Investigational Site, Mainz
  - 1307.4.49001 Boehringer Ingelheim Investigational Site, Neuss